CLINICAL TRIAL: NCT02927002
Title: Effects of Non-invasive Brain on Decision-making in Impulse Control Disorders
Brief Title: Effects of Non-invasive Brain Stimulation in Impulse Control Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2014-374
Record Dates: First submitted 2016-05-17; First posted 2016-10-06 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Impulse Control Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noninvasive brain stimulation: active (Active Comparator): In active condition, subject will receive stimulation during all the 30-minute stimulation period
  Interventions: Device: Noninvasive brain stimulation
- Noninvasive brain: sham (Sham Comparator): In sham condition, subject will receive stimulation only at the beginning and at the end of 30-minute stimulation period.
  Interventions: Device: Noninvasive brain stimulation

INTERVENTIONS:
Device: Noninvasive brain stimulation

SUMMARY:
The goal of this project is to study the effect of noninvasive brain stimulation on decision-making and on brain activity in impulse control disorders.

ELIGIBILITY:
Inclusion Criteria:

* Impulse control disorders according to DSM-IV criteria

Exclusion Criteria:

* Other psychiatric disorders
* Contraindication to Non-invasive brain stimulation and MRI

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Change in decision-making from pre to post stimulation assessed with the Balloon Analogue Risk Task | 10 minutes before and immediately after the 30 minutes of non invasive brain stimulation

SECONDARY OUTCOMES:
Changes in brain activity assessed between before and during stimulation measured with functional magnetic resonance (fMRI) | 20 minutes before and immediately after the 30 minutes of non invasive brain stimulation
Neural metabolites concentrations measured with magnetic resonance spectroscopy (MRS) | 20 minutes before and immediately after the 30 minutes of non invasive brain stimulation
Change in Craving from pre to post stimulation assessed with a single standardized scale | 7 minutes before and 3 minutes after the end of the 30 minutes of non invasive brain stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Interdisciplinaire de Recherche en Réadaptation et Intégration, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided